CLINICAL TRIAL: NCT03100422
Title: Strategies of Therapy With the Exoskeleton Robot ARMinMulti VIT-ARMin
Brief Title: Strategies of Therapy With the Exoskeleton Robot ARMin
Acronym: MultiVIT-ARMin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Rehaklinik Zihlschlacht AG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Multi VIT-ARMin
Record Dates: First submitted 2017-02-14; First posted 2017-04-04 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: randomized
Who Masked: Investigator, Outcomes Assessor
Masking Description: Lots will be drawn that assign to either robotic therapy or occupational therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARMin (Experimental): Therapy with the arm therapy robot ARMin
  Interventions: Device: ARMin
- Arm+ occupational therapy (Active Comparator): a form of conventional occupational therapy that involves both arms
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Device: ARMin — arm therapy robot
  Arms: ARMin
Other: Occupational Therapy — bilateral arm training
  Arms: Arm+ occupational therapy

SUMMARY:
Neurological patients (e.g., after stroke) need long-term neurorehabilitation therapy of the arm with often limited, unsatisfactory outcome. Robots became a promising supplement or even alternative for neurorehabilitation training.

DETAILED DESCRIPTION:
The exoskeleton robot ARMin was further developed and software components adapted accordingly to offer a unique intensified and patient-tailored robot-aided training of the arm. The goal is to enhance treatment efficacy to an extent that the improvement in motor function is meaningful for the individual patient. The study objective is to compare ARMin therapy and a form of conventional occupational therapy that involves both arms regarding change in motor function.

ELIGIBILITY:
Inclusion Criteria:

* - Aged ≥18 years
* Ischemic cerebral vascular accident (CVA, stroke) in the sub-acute phase (one to twelve weeks post-stroke) as verified by brain imaging (CT or MRI)
* Inpatient at Rehaklinik Zihlschlacht, Switzerland
* Decreased arm motor function in one arm with a FMA of 8 to 20 points (out of 66)
* No excessive spasticity of the affected arm (modified Ashworth Scale mAS ≤3) as assessed by the physician
* No serious medical or psychiatric disorder as assessed by the physician
* No serious orthopaedic, rheumatologic or other disease restricting movements of the paretic arm as assessed by the physician
* No clinically significant shoulder subluxation (palpation <2 fingers) as assessed by the physician
* No skin ulcerations at the paretic arm as assessed by the physician
* Ability to communicate effectively with the examiner such that the validity of the patient's data could not be compromised as assessed by the physician
* No history of cyber sickness (e.g., nausea when looking at a screen or playing computer games) as assessed by the physician
* No pacemaker or other implanted electric device as verified by patient record
* Bodyweight <120 kg
* No serious cognitive defects or aphasia preventing effective use of ARMin as assessed by the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment, upper extremity motor function | from baseline to day 3 post-training
  impairment based clinical test

SECONDARY OUTCOMES:
ARMin assessment time | from baseline to day 3 post-training
  time
ARMin assessment torques | from baseline to day 3 post-training
  torques
ARMin assessment positions | from baseline to day 3 post-training
  positions
Intrinsic Motivation Inventory | from baseline to day 3 post-training
  questionnaire
Motor Activity Log | from baseline to day 3 post-training
  questionnaire
handheld dynamometer | from baseline to day 3 post-training
  isometric strength

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, PhD, Principal Investigator — ETH Zurich
Locations (1):
- Labor für Sensomotorische Systeme, ETH Zürich, Balgrist Campus, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided